CLINICAL TRIAL: NCT01057901
Title: 24 - Week Flibanserin 100mg for the Treatment of Hypoactive Sexual Desire Disorder in Postmenopausal Women in Noth America
Brief Title: Flibanserin for the Treatment of Hypoactive Sexual Desire Disorder in Postmenopausal Women in North America
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated for administrative reasons.
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.156
Record Dates: First submitted 2010-01-25; First posted 2010-01-28 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flibanserin 100 mg (Experimental): Flibanserin 100 mg administered at bedtime
  Interventions: Drug: Flibanserin
- Placebo (Placebo Comparator): This is the matched placebo which will be administered two tablets daily at bedtime.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flibanserin — Flibanserin 100mg administered at bedtime for 24 weeks
  Arms: Flibanserin 100 mg
Drug: Placebo — This is the matched placebo which will be administered two tablets daily at bedtime.
  Arms: Placebo

SUMMARY:
The objective of this trial is to assess the safety and efficacy of 24-week course of flibanserin for the treatment of Hypoactive Sexual Desire Disorder (HSDD) in naturally postmenopausal women.

ELIGIBILITY:
Inclusion criteria:

* Naturally postmenopausal women of any age with at least one ovary
* Diagnosis of Hypoactive Sexual Desire Disorder, generalized acquired type,of at least six months duration
* Stable, monogamous heterosexual relationship for at least one year
* Willing to discuss sexual issues
* Willing to engage in sexual activity at least once a month
* Normal Pap smear
* Normal mammogram
* Normal uterine lining
* Able to comply with daily use of handheld data entry device

Exclusion criteria:

* Sexual dysfunctions other than HSDD, such as Sexual Aversion Disorder, Substance-induced Sexual Dysfunction, Dyspareunia, Vaginismus, Gender Identity Disorder, Paraphilia and Sexual Dysfunction due to a General Medical Condition
* Partner with inadequately treated organic or psychosexual dysfunction
* Sexual function impaired by psychiatric disorder
* Sexual function impaired by gynecological disorder
* Major Depression
* Suicidal behavior or ideation
* Major life stress that could impair sexual function
* Substance abuse

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (100):
- United States (84):
  - 511.156.01059 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.156.01084 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 511.156.01053 Boehringer Ingelheim Investigational Site, Tuscon, Arizona
  - 511.156.01069 Boehringer Ingelheim Investigational Site, Tuscon, Arizona
  - 511.156.01063 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 511.156.01076 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 511.156.01039 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 511.156.01070 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 511.156.01075 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 511.156.01087 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 511.156.01064 Boehringer Ingelheim Investigational Site, Newport Beach, California
  - 511.156.01016 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 511.156.01007 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.156.01038 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.156.01067 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 511.156.01036 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.156.01092 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 511.156.01027 Boehringer Ingelheim Investigational Site, New London, Connecticut
  - 511.156.01022 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 511.156.01042 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 511.156.01047 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 511.156.01051 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 511.156.01011 Boehringer Ingelheim Investigational Site, Gainseville, Florida
  - 511.156.01078 Boehringer Ingelheim Investigational Site, Lake Worth, Florida
  - 511.156.01095 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.156.01046 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 511.156.01056 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 511.156.01045 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 511.156.01021 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 511.156.01081 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 511.156.01066 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 511.156.01025 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.156.01028 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.156.01089 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 511.156.01010 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 511.156.01008 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 511.156.01034 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 511.156.01012 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 511.156.01074 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 511.156.01079 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 511.156.01080 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 511.156.01006 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 511.156.01086 Boehringer Ingelheim Investigational Site, Paw Paw, Michigan
  - 511.156.01005 Boehringer Ingelheim Investigational Site, Chaska, Minnesota
  - 511.156.01013 Boehringer Ingelheim Investigational Site, Olive Branch, Mississippi
  - 511.156.01088 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.156.01001 Boehringer Ingelheim Investigational Site, New Brunswick, New Jersey
  - 511.156.01055 Boehringer Ingelheim Investigational Site, Plainsboro, New Jersey
  - 511.156.01037 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 511.156.01031 Boehringer Ingelheim Investigational Site, Purchase, New York
  - 511.156.01009 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 511.156.01024 Boehringer Ingelheim Investigational Site, Cary, North Carolina
  - 511.156.01065 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 511.156.01029 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 511.156.01002 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 511.156.01040 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 511.156.01026 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.156.01093 Boehringer Ingelheim Investigational Site, Bismarck, North Dakota
  - 511.156.01052 Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - 511.156.01017 Boehringer Ingelheim Investigational Site, Beachwood, Ohio
  - 511.156.01032 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.156.01033 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.156.01068 Boehringer Ingelheim Investigational Site, Englewood, Ohio
  - 511.156.01077 Boehringer Ingelheim Investigational Site, Ashland, Oregon
  - 511.156.01072 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 511.156.01082 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 511.156.01094 Boehringer Ingelheim Investigational Site, West Reading, Pennsylvania
  - 511.156.01083 Boehringer Ingelheim Investigational Site, Warwick, Rhode Island
  - 511.156.01048 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 511.156.01058 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 511.156.01085 Boehringer Ingelheim Investigational Site, Watertown, South Dakota
  - 511.156.01073 Boehringer Ingelheim Investigational Site, Bristol, Tennessee
  - 511.156.01041 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 511.156.01035 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 511.156.01091 Boehringer Ingelheim Investigational Site, Jackson, Tennessee
  - 511.156.01060 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 511.156.01003 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 511.156.01054 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 511.156.01050 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 511.156.01014 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.156.01049 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.156.01015 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.156.01090 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.156.01020 Boehringer Ingelheim Investigational Site, Seattle, Washington
- Canada (16):
  - 511.156.02004 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 511.156.02010 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 511.156.02009 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 511.156.02014 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 511.156.02012 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 511.156.02017 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 511.156.02007 Boehringer Ingelheim Investigational Site, Woodstock, New Brunswick
  - 511.156.02008 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 511.156.02001 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 511.156.02013 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 511.156.02006 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 511.156.02005 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.156.02016 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 511.156.02002 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 511.156.02015 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 511.156.02003 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Portman DJ, Brown L, Yuan J, Kissling R, Kingsberg SA. Flibanserin in Postmenopausal Women With Hypoactive Sexual Desire Disorder: Results of the PLUMERIA Study. J Sex Med. 2017 Jun;14(6):834-842. doi: 10.1016/j.jsxm.2017.03.258. PMID 28583342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flibanserin 100 mg | Placebo
Started | 376 | 372
Completed | 116 | 126
Not Completed | 260 | 246

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin 100 mg | Placebo | Total
Number analyzed (Participants) | 376 | 372 | 748
Age, Customized [Number; unit: participants]
  less than 45 years | 4 | 5 | 9
  45-54 years | 154 | 128 | 282
  55-64 | 196 | 212 | 408
  65 years and older | 22 | 27 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 376 | 372 | 748
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 324 | 310 | 634
  White Hispanic | 18 | 27 | 45
  Black/African American | 25 | 26 | 51
  Black/African American Hispanic | 1 | 1 | 2
  Asian | 8 | 4 | 12
  Asian Hispanic | 0 | 0 | 0
  American Indian/Alaskan Native | 0 | 2 | 2
  Hawaiian/Pacific Islander | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Satisfying Sexual Events
Description: The change from baseline in the number of SSE's as measured by the eDiary. The calculation of Satisfying Sexual Event (SSEs) will be standardized to a 28-day period according to the below formula:
  Total monthly events = 28 x (sum of the number of events) / (sum of number of days entered).
  "Satisfying" means gratifying, fulfilling, satisfactory, and/or successful for the patient. The partner's satisfaction is not the subject of this question.
Time Frame: baseline to 24 weeks
Population: The full analysis set (FAS), consisted of those patients who were randomized to a treatment group, received at least one dose of study medication, had at least one baseline value of either one of the co-primary endpoints or key secondary endpoint, and had usable data.
Measure: Mean (Standard Deviation); unit: SSEs/month
Arm/Group | Flibanserin 100 mg | Placebo
Number analyzed (Participants) | 346 | 335
SSEs/month | 1.0 (3.3) | 0.7 (2.9)

2. Primary Outcome: Change From Baseline in the Score on the Female Sexual Function Index (FSFI) Desire Domain
Description: The Female Sexual Function Index (FSFI) is a brief, multidimensional, self-administered questionnaire for assessing key domains of sexual function in women. The scale consists of 19 items that assess sexual function over the past four weeks and yields scores in six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The two items in the desire domain are scored from 1 to 5 (1 is lowest level of desire and 5 is the highest level of desire). The raw scores of the two items are added together and then multiplied by the domain factor of 0.6. Thus, the score of the desire domain ranges from 1.2 (lowest level of desire) to 6.0 (highest level of desire). For the entire instrument, each of the six domains contributes a maximum of 6 points to the total. Scores on the full scale range from a minimum of 2 to a maximum of 36.
Time Frame: baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flibanserin 100 mg | Placebo
Number analyzed (Participants) | 351 | 343
units on a scale | 0.6 (0.1) | 0.4 (0.1)

ADVERSE EVENTS:
Description: Among the 372 randomized patients, 369 took at least one dose of study medication and had at least one post-dose on-treatment safety assessment. These patients were included in the treated set that was analyzed for safety.
Arm/Group | Flibanserin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/376 | 4/369
Other Adverse Events (participants affected / at risk) | 118/376 | 74/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100 mg (N=376) | Placebo (N=369)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Breast Cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischemic event (Nervous system disorders) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100 mg (N=376) | Placebo (N=369)
Insomnia (Psychiatric disorders) | 29 (30) | 14 (14)
somnolence (Nervous system disorders) | 26 (27) | 8 (9)
headache (Nervous system disorders) | 19 (21) | 24 (27)
dizziness (Nervous system disorders) | 24 (28) | 13 (14)
nausea (Gastrointestinal disorders) | 20 (21) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No